CLINICAL TRIAL: NCT06257810
Title: Impact of Differential and Systematic Dengue, Chikungunya, and Malaria Diagnostics on Patient Management and Antibiotic Use in Burkina Faso and Ivory Coast
Brief Title: Impact of Differential and Systematic Diagnosis of Dengue, Chikungunya and Malaria on Patient Management and Antibiotic Use in West Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E0545
Record Dates: First submitted 2023-11-27; First posted 2024-02-14 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Dengue; Chikungunya; Malaria
Keywords: Diagnosis; Clinical Management; Antibiotic; Patient Management; Immunoassays; Arboviruses; West Africa; Antibiotic resistance; Dengue; Malaria; Chikungunya
MeSH Terms: conditions — Dengue; Chikungunya Fever; Malaria; Disease

STUDY DESIGN:
Intervention Model Description: This is a multicentric study which will be carried out in four hospitals, two in Burkina Faso and two in Ivory Coast. In each of these two countries, an "intervention" site and a "control" site will be included in the study. The study is interventional as the investigators collected additional blood samples than the routine practices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Site (Active Comparator): In the interventional sites, bioMérieux teams provided training to raise awareness of the diagnosis of dengue, chikungunya and malaria. In addition, a VIDAS instrument was installed and dengue and chikungunya diagnostic kits were supplied so that diagnosis could be carried out systematically for each patient included.
  Interventions: Diagnostic Test: VIDAS® Dengue Antigen NS1, VIDAS® Anti-Dengue IgM, VIDAS® Anti-Dengue IgG, VIDAS® Anti-Chikungunya IgM and VIDAS® Anti-Chikungunya IgG
- Control Site (Placebo Comparator): In the control centres, only routine practices were observed.
  Interventions: Other: Standard of care practices

INTERVENTIONS:
Diagnostic Test: VIDAS® Dengue Antigen NS1, VIDAS® Anti-Dengue IgM, VIDAS® Anti-Dengue IgG, VIDAS® Anti-Chikungunya IgM and VIDAS® Anti-Chikungunya IgG — For patients managed in an "intervention site", a diagnostic test for dengue and chikungunya using VIDAS® as well as a screening test for malaria will be carried out. An awareness campaign on the use of VIDAS® diagnostic tests will be implemented as well.
  The diagnosis will be based on the patient's clinical symptoms, the biological results of the VIDAS® tests for dengue and chikungunya, as well as the results of the tests for malaria.
  Arms: Intervention Site
Other: Standard of care practices — For patients managed in a "control site", the standard of care practices will be applied in the case of a febrile condition of undetermined etiology. This includes clinical diagnosis and, where appropriate, the use of routinely available diagnostic tests. At the end of the study, the collected samples will be tested using VIDAS® differential diagnosis tests to estimate the number of cases of dengue and chikungunya that have not been correctly diagnosed.
  Arms: Control Site

SUMMARY:
The differential and systematic diagnosis of malaria, dengue and chikungunya in patients with fever (≥38.5°C) of undetermined etiology would allow the identification of infection by these pathogens and thus limit the inappropriate use of antibiotics (discontinuation or non-initiation) and optimize the clinical management and prognosis of patients.

DETAILED DESCRIPTION:
The research hypotheses are as follows:

* Systematic diagnosis of malaria, dengue and chikungunya using diagnostic tests would improve the clinical management of patients with fever of undetermined etiology and reduce the misuse of antibiotics (discontinuation or non-initiation) and associated resistance.
* Improved management is associated with a reduction in the use of hospital resources, professional inactivity and an improvement in the quality of life and satisfaction of patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years
* Patient with fever (≥38.5°C) and at least two of the following symptoms in the last 10 days:

  * Severe headache
  * Retro-orbital pain
  * Muscle and joint pain
  * Nausea
  * Vomiting
  * Adenopathy
  * Rash
  * Abdominal pain
  * Asthenia
  * Spontaneous bleeding (purpura, epistaxis, haematemesis, etc)
* Willingness and ability to provide two 4 mL blood samples
* Willingness to provide one drop of blood per capillary sample
* Informed and signed consent

Exclusion Criteria:

* Subjects aged < 18 years
* Pregnant women
* Breastfeeding women
* Patient's refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Rate of antibiotic prescription | Inclusion and Day 7
  Rate of antibiotic prescription (discontinuation or non-initiation).

SECONDARY OUTCOMES:
Consumption of hospital resources | Day 7
  Number of days in hospital.
Consumption of hospital resources | Day 7
  Number of hospital visits within 7 days.
Patient satisfaction | Inclusion and Day 7
  Patient satisfaction with the health care (measured on a scale of 1 (worse) to 5 (better)).
Patient's quality of life | Inclusion and Day 7
  Percentage on patient's quality of life (1 (worse) to 100 (better)) + EQ-5D questionnaire.
Patient's loss of productivity | Inclusion and Day 7
  Questionnaire on number of working day lost.

OTHER OUTCOMES:
Prevalence of dengue, chikungunya and malaria | Inclusion, after lab results (an average of one day)
  To determine the prevalence of dengue, chikungunya and malaria in patients with fever (≥38.5°C) of undetermined etiology
Clinical situations associated with inappropriate antibiotic prescription | Inclusion and Day 7
  Number of clinical situations associated with inappropriate antibiotic prescription, including suggestive signs of bacterial infection or severe sepsis such as neurological, cardio-circulatory failure, coma or purpura fulminans
Rate of antibiotic prescription | Up to 7 days
  To estimate the impact of differential diagnosis testing on the rate of antibiotic prescription in patients with dengue and/or chikungunya

CONTACTS AND LOCATIONS:
Locations (3):
- Institut de Recherche en Sciences de la Santé, Ouagadougou, Burkina Faso
- Côte d’Ivoire (2):
  - CHU Cocody, Abidjan, Cocody
  - CHU Treichville, Abidjan, Treichville

IPD SHARING:
Plan to Share IPD: No